CLINICAL TRIAL: NCT03404128
Title: Long Term Follow-up of Patients Treated With Hippocampal Deep Brain Stimulation for Refractory Epilepsy
Brief Title: Long Term Follow-up of Hippocampal DBS for Refractory Epilepsy
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Neurologie, Principal Investigator (Prof. dr. Paul Boon), University Hospital, Ghent
Other Study IDs: LT FU HC-DBS
Record Dates: First submitted 2017-12-01; First posted 2018-01-19 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Refractory Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaires: Questionnaire for patient Questionnaire for neurologist
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Questionnaire for patient: satisfaction regarding rechargeable DBS battery Questionnaire for neurologist: seizure frequency, satisfaction regarding rechargeable DBS battery

SUMMARY:
Follow up of the patients at Ghent University Hospital treated with hippocampal DBS for refractory epilepsy.

Endpoints:

* Long term evaluation of the effects of hippocampal DBS on seizure frequency and cognition
* Evaluation of the satisfaction of patients and neurologist regarding the rechargeable DBS battery

ELIGIBILITY:
Inclusion Criteria:

* Treated with hippocampal DBS for refractory epilepsy at Ghent University Hospital

Exclusion Criteria:

* (none)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with refractory epilepsy treated with hippocampal DBS
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Seizure frequency per month based on seizure diary | Every six months (up to 2 years after implantation of rechargeable device)
  Efficacy measured by reduction in seizure frequency before and after implantation

SECONDARY OUTCOMES:
Cognition | Yearly (up to 2 years after implantation of rechargeable device)
  Cognition measured by neuropsychological testing
Number of device problems | Every six months (up to 2 years after implantation of rechargeable device)
  Reporting of device problems including long charging time, bad connection between device and charger, high frequency of charging (> 1 time a day).
Number of adverse events | Every six months (up to 2 years after implantation of rechargeable device)
  Reporting of adverse events after implantation

CONTACTS AND LOCATIONS:
Overall Officials: Paul Boon, MD, PhD, Principal Investigator — UZ Gent

IPD SHARING:
Plan to Share IPD: Undecided